CLINICAL TRIAL: NCT06950944
Title: Efficacy and Safety of Repeated-use Middle Cut Off Membrane Dialyzers on Middle Molecule Uremic Toxin and Inflammatory Cytokine Clearances in Hemodialysis Patients
Brief Title: Efficacy and Safety of Repeated-use Middle Cut Off Membrane Dialyzers in Hemodialysis Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Eakalak Lukkanalikitkul, Principal Investigator, Nephrologist, Khon Kaen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HE661417
Record Dates: First submitted 2024-02-06; First posted 2025-04-30 (Actual); Last update posted 2025-05-04 (Actual); Status verified 2025-04

CONDITIONS: Hemodialysis; Hemodialysis Treatment; Dialysis Adequacy
Keywords: Middle cutoff membrane dialyzer; Uremic toxin clearance; Reused membrane dialyzer

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Theranova 500 (Experimental): The participant underwent dialysis using the Theranova 500 dialyzer
  Interventions: Device: Theranova 500
- Elisio 21Hx (Active Comparator): The participant underwent dialysis using the Elisio 21Hx dialyzer
  Interventions: Device: Theranova 500

INTERVENTIONS:
Device: Theranova 500 — Participants will dialysis by Theranova 500 dialyzer during study period, the dialyzer will reprocessing with standard hospital protocol and dialyzer will check before use in dialysis session.

SUMMARY:
The goal of this clinical trial is to compare the efficacy of uremic toxin and inflammatory cytokine clearance by using reprocessing middle cutoff membrane (MCO) dialyzer in chronic hemodialysis patients. The main questions it aims to answer are:

* To evaluate efficacy of uremic toxin and inflammatory cytokine clearance and safty of hemodialysis with reprocessing MCO dialyzer compared with new MCO dialyzer
* To compare efficacy of uremic toxin and inflammatory cytokine clearance between 2 types of MCO dialyzer which availble in Thailand (Theranova 500 and Elisio 21Hx).

Participants will randomized to 2 types of MCO groups after that they will receive hemodialysis by using study dialyzer with similar hemodialysis prescription. The dialyzer in this study were reprocessing by standard hospital protocol. Researchers will compare 2 types of dialyzer groups to see efficacy of uremic toxin and inflammatory cytokine clearance and safety of use reprocessing dialyzer.

DETAILED DESCRIPTION:
Study design and population The single - center prospective open-label randomize control trial was conducted in prevalence HD patients at the Srinagarind Hospital, Khon Kaen University between January 2024 and March 2024. The inclusion criteria were participants aged 18-80 years old, with adequate HD (spKt/V > 1.2 and 1.8 per session for patients undergoing thrice- and twice-weekly HD, respectively) for more than 3 months, utilizing arteriovenous fistula or graft (AVF or AVG) for vascular access. The exclusion criteria were pregnancy, vascular access dysfunction, contraindicated to reprocess dialyzer (e.g., blood-transmitted infections such as HBV, HIV, and MDR pathogens), advanced-stage cancer or cardiovascular diseases, severe comorbidities with less than a 1-year life expectancy, prior severe infections or hospitalization within 3 months or receiving immunosuppressive drugs, and history of severe dialyzer allergy.

Study Intervention All enrolled 48 participants were randomized to hemodialysis using Theranova 500 dialyzer or Elisio 21HX dialyzer stratified by age, sex, causes of ESRD, dialysis vintage, dialysis sessions per week and type of vascular accesses.Each patient received twice and thrice weekly 4-hour dialysis sessions with their usual prescriptions including blood and dialysate flow rates, dialysate composition, intradialytic coagulant and dry weight. Both groups utilizing the Fresenius 4008H machine for dialysis treatment, with the study concluding when complete of 15th dialysis session or study dialyzer was disqualified for reused adhering to the standard dialyzer reprocessing protocol in Srinagarind hospital. Intradialytic monitoring and treatment of intradialytic complications were performed by trained HD nurses. The ultrapure quality dialysis water defined by total microbial counts < 0.1 CFU/mL and endotoxin concentrations < 0.03 EU/mL was used in both groups. Both study dialyzers underwent disinfection with 2% peracetic acid and reprocessed using an automatic dialyzer reprocessing machine. In cases where abnormalities or blood clots were detected by the automatic machine, trained staff conducted a reassessment and rinsed the dialyzer with reverse osmosis water until the clot dissipated. The dialyzers exhibiting a reduction TCV exceeding 20% or unable to clear blood clots were deemed unsuitable for reprocessing and were disposed.

Data collection and definition of outcomes Baseline characteristics and demographic data, e.g., age, sex, weight, height, body mass index, comorbid diseases, causes of ESKD, physical status, and socioeconomic data were collected from the interview, physical examination, and review of medical records. Baseline laboratory data were collected 2-week prior to the study period. The efficacy of various-size uremic toxins removal including phosphorus, urea, creatinine, homocysteine, PTH, β2-MG, κ-FLC and λ-FLC together with inflammatory markers including IL-6 and C-reactive protein (CRP) were evaluated by pre- to post-dialysis RRs at 1st, 2nd, 5th, 10th, 15th session of dialysis intervention. The RR was calculated by the following equations according to Bergström and Wehle. Techniques for measurement of serum solute levels composed of molecular absorption spectrometry (for urea and creatinine), immunoturbidimetric assay (for β2-MG and CRP), electrochemiluminescence immunoassay (for IL-6), enzymatic assay (for homocysteine), and latex particle enhance immunoturbidimetric method (for κ-FLC and λ-FLC). Regarding of safety outcomes, data of dialyzer related complications including dialyzer reaction, rupture of dialyzer membranes, and intradialytic dialyzer clot were collected.

ELIGIBILITY:
Inclusion Criteria:

* chronic hemodialysis with dialysis vintage more than 3 months
* hemodialysis via permanent vascular access (fistula or graft)
* adequate hemodialysis define with spKt/V > 1.8 and > 1.2 per session in twice and thrice weekly hemodialysis, respectively

Exclusion Criteria:

* preganancy
* hemodialysis vascular access dysfunction
* blood transmitted infection
* advanced malignancy or severe morbidity with life expectancy less than 1 year
* severe dialyzer reaction
* receive immunosuppressive drug

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Efficacy of uremic toxin clearances from repeated-use middle cut off membrane dialyzers | up to 3 months or 12 weeks
  The efficacy of various-size uremic toxins removal including phosphorus, urea, creatinine, homocysteine, PTH, β2-MG, κ-FLC and λ-FLC together with inflammatory markers including IL-6 and C-reactive protein (CRP) were evaluated by pre- to post-dialysis reduction ratio (RRs) at 1st, 2nd, 5th, 10th, 15th session of dialysis intervention. The RR was calculated by the following equations according to Bergström and Wehle.

SECONDARY OUTCOMES:
Albumin loss from hemodialysis | up to 3 months or 12 weeks
  The loss of albumin from dialysis was calculated from area under the dialysate albumin concentration-time curve (AUC) of measurement of albumin quantity in the dialysis fluid at initial, 60, 120 min and at the end of dialysis sessions.
Adveres event from reused middle cutoff membrane dialyzer | up to 3 months or 12 weeks
  Data of dialyzer related complications including, intradialytic hypotension (nadir systolic blood pressure less than 90 mmHG or drop from predialysis more than 40 mmHg), dialyzer reaction, rupture of dialyzer membranes, and intradialytic dialyzer clot were collected.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Khon Kaen University, Khon Kaen, Changwat Khon Kaen, Thailand

IPD SHARING:
Plan to Share IPD: No